CLINICAL TRIAL: NCT03261167
Title: A Phase III Study (a Placebo Controlled, Randomized, Double-blind Comparative Study and an Open-label, Uncontrolled Study) to Evaluate the Efficacy and Safety of GSK1358820 in Patients With Post-stroke Upper Limb Spasticity
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of GSK1358820 in Subjects With Post-stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207660
Record Dates: First submitted 2017-08-23; First posted 2017-08-24 (Actual); Results first posted 2019-10-18 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Spasticity, Post-Stroke
Keywords: Botulinum toxin A; Safety; post-stroke upper limb spasticity; Efficacy; GSK1358820; double blind
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Subjects will receive either 400 units of botulinum toxin A injection or 240 units of botulinum toxin A injection plus placebo in double blind phase. Eligible subjects for open-label treatment period will receive 400 units of botulinum toxin A injection.
Who Masked: Participant, Investigator
Masking Description: This study will contain a double blind treatment period (Part 1) followed by open-label treatment period (Part 2/Part3/Part4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Subjects receiving 400 units of botulinum toxin A (Experimental): Subjects will receive a total dose of 400 units of botulinum toxin A of which 240 units will be injected into the muscles that act on finger (including thumb flexors) and wrist flexors, and a total of 160 units will be injected into the muscles that act on the elbow flexors.
  Interventions: Drug: Botulinum toxin A (GSK1358820)
- Part 1: Subjects receiving 240 units of botulinum toxin A (Active Comparator): Subjects will receive 240 units of botulinum toxin A injected into the muscles that act on the finger (including thumb flexors) and wrist flexors. Placebo will be injected into the muscles that act on the elbow flexors.
  Interventions: Drug: Botulinum toxin A (GSK1358820); Drug: Placebo
- Part 2,3,4: Subjects receiving 400 units of botulinum toxin A (Experimental): Subjects will receive botulinum toxin A with a dose of 400 units injected in a divided doses.
  Interventions: Drug: Botulinum toxin A (GSK1358820)

INTERVENTIONS:
Drug: Botulinum toxin A (GSK1358820) — GSK1358820 is sterile, purified type A botulinum neurotoxin complex. GSK1358820 injection will contain botulinum toxin A (100 units), sodium chloride (0.9 milligrams [mg]), and human serum albumin (0.5 mg). It will be available with doses of 400 units and 240 units.
Drug: Placebo — Placebo injection will contain sodium chloride (0.9 mg).
  Arms: Part 1: Subjects receiving 240 units of botulinum toxin A

SUMMARY:
Botulinum toxin A (GSK1358820) is a sterile, purified type A botulinum neurotoxin complex. In Japan, 240 units of botulinum toxin A are approved as a maximum dose per administration for upper limb spasticity. This study is planned to evaluate the effectiveness and safety of 400 units of botulinum toxin A which can help to increase the maximum dose per administration to 400 units from 240 units as the treatment with 240 units is considered insufficient in subjects with post-stroke upper limb spasticity. Approximately 120 subjects will be randomized to receive either 400 or 240 units of botulinum toxin A in double blind phase followed by open-label phase in which 400 units of the study treatment will be injected in both the groups. The study period will be up to 52 weeks, consisting of a screening phase up to 4 weeks, minimum 12-week double blind phase (Part 1), maximum 36- week open-label phase (12 weeks per cycle with 3 treatment phases: Part 2, Part 3 and Part 4).

ELIGIBILITY:
Inclusion Criteria:

* For screening phase (Day -28 to Day -1): Between 20 and 80 years of age at the time of informed consent (ICF).
* Subjects with at least a 3-month history of upper limb spasticity after the most recent stroke.
* Subjects who have spastic symptoms in the finger (including the thumb), wrist, and elbow flexors whom the investigator considers the injections of 400 units of the product is necessary for the upper limb based on the muscle spasms and the symptoms of the subject.
* Subjects who have a previous treatment history of 240 units of the product for the upper limb at least 16 weeks before screening.
* Subjects who meet following criteria on MAS at screening (Test position : sitting): at least 3 in for the elbow flexors and at least 2 in the finger or wrist flexors.
* Subjects who have severe upper limb spasticity, which deserves to be treated with 400 units of the product in the divided dose and was previously injected 240 units of the product.
* Subjects whom the investigator considers that enrolment in the study poses no problems based on the laboratory data results at screening.
* Subjects who are free from a history of acute decreased lung function (hospitalization with aggravated asthma/ chronic obstructive pulmonary disease (COPD), pneumonia, or signs of pneumonia, or abnormal reactive airway diseases suggested on X-rays) within the last 3 months at screening and have stable pulmonary function (oxygen saturation [SpO2]value is >=95%).
* Body weight >=40 kilograms (kg) at screening.
* Male or female subjects will be included. Male subjects must content to use highly effective contraceptive methods and sperm donation must be avoided. Female subjects who are not pregnant or lactating are considered eligible if at least one of the following criteria is met; non-childbearing potential, women of childbearing potential who content to follow the guidance about contraception during the study period and at least for 3 months after the last dose of the product, no plan of pregnancy during the study period.
* Subjects who have ability to sign their name on the ICF.
* For enrolment in the study (Day 1 [prior to injection]):Subjects who meet the following criteria on MAS score: (Test position : sitting): At least 3 in the elbow flexors and at least 2 in the finger or wrist flexors.
* If centrally acting muscle relaxants, tetracycline antibiotics, anticholinergics, benzodiazepines, or benzamides are given, the dose and regimen must be stable at least for the last 2 months before Day 1; Subjects who can maintain the same dosage and regimens at least in the blind phase after initial injection (dose reductions and discontinuation of the drugs are acceptable in the open-label phase. However, second dose increase, resumption, and or new treatment will not be performed).
* If intrathecal baclofen is given, the dose and regimen must be stable at least for the last 1 month before Day 1; Subjects who can maintain the same dosage and regimens at least in the blind phase after initial injection (intravenous bolus is not acceptable, dose reductions and discontinuation of the drugs are acceptable. However, second dose increase, resumption, and or new treatment will not be performed).
* If antiepileptic agents are given, the dose and regimen must be stable at least for the 1 month before Day 1; Subjects who can maintain the same dose and regimens at least in the blind phase after initial injection (dose reductions and discontinuation of the drugs are acceptable in the open-label phase. However, second dose increase, resumption, and new treatment will not be performed).
* If a physical therapy, occupational therapy, or a static splint on the study involvement upper limbs is given, the frequency and treatment regimen must be stable at least for the last 3 weeks before Day 1; Subjects who can maintain the same dose and regimens at least in blind phase (In the open-label phase, the frequency and treatment regimen can be changed depending on the condition of spasticity).

Exclusion Criteria:

* For screening phase (Day -28 to Day -1): Subjects present with spasticity requiring treatment in the non-paralytic side of the upper limb.
* Subjects who have fixed contracture in the finger (upper limb), wrist, elbow or shoulder muscle, which will be involved in the study.
* Subjects who have medically significant capsulitis or subluxation in any one of the fingers (upper limb), wrist, elbow and shoulder, which will be involved in the study, or whom a investigator considers the complicated local signs of pain may affect the efficacy evaluation.
* Subjects's upper limb spasticity is attributed to other than stroke (traumatic brain injury, spinal cord injury, multiple sclerosis, or cerebral palsy).
* Subjects who have a 2-fold higher alanine aminotransferase (ALT) level than the upper limit of normal (ULN).
* Subjects who have a 1.5-fold higher bilirubin than the ULN (If a bilirubin fractionation shows direct bilirubin < 35%, a 1.5-fold higher free bilirubin than the ULN is acceptable).
* Subjects whom the investigator considers presence of a current medical history of unstable liver diseases or biliary tract diseases (the condition will be defined by development of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice or hepatic cirrhosis).
* Subjects with corrected QT interval (QTc) > 450 milliseconds (msec) or QTc > 480 msec in subjects with bundle branch block.
* Subjects who use peripherally acting muscle relaxants (dantrolene sodium, suxamethonium chloride, pancuronium bromide, vecuronium bromide, rocuronium bromide, etc.) within 1 week of screening.
* Subjects who use antibiotic agents with neuromuscular junction inhibitory effects: Aminoglycoside antibiotic agents (streptomycin sulfate, kanamycin sulfate, gentamicin sulfate, neomycin sulfate, spectinomycin hydrochloride, etc.), polypeptides (polymyxin B sulfate), lincomycins (lincomycin hydrochloride, clindamycin), and enviomycin sulfate within 1 week of screening.
* Subjects who was diagnosed as having a malignant tumor, or have a history of a malignant tumor within the last 5 years (except completely resected basal cell carcinoma or planocellular carcinoma at least 12 weeks before screening).
* Subjects who have participated in another study of an investigational product or other medical research (a clinical study of pharmacotherapy, non-pharmacotherapy, or interventional device) within 30 days before screening, or are currently participating in a study.
* Subjects who are concerned likely to have an increased risk for an underlying medical condition/neurological disease due to exposure of the product; subjects who have myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or a serious disease and use of a concomitant drug which may inhibit neuromuscular function.
* Subjects with antihuman immunodeficiency virus (HIV) antibody positive.
* Subjects who previously experienced allergic reactions or hypersensitivity due to botulinum toxin type A, an additive agent of sodium chloride, or human serum albumin.
* Subjects who were previously suspected to have neutralizing antibody production by a investigator during an injection of botulinum toxin type A.
* Subjects who have a skin disease such as infection at the site to be injected.
* Subjects who suffer from serious and unstable disease, which could pose problems for the safety of subjects and study procedure compliance.
* For enrolment in the study (Day 1 [prior to injection]): Subjects who have aspiration pneumonia, relapse of lower respiratory tract infection, uncontrollable asthma, uncontrollable COPD, and/or underlying or a history of serious respiratory dysfunction, which were clinically considered to be respiratory function impairment by a investigator within 12 months before Day 1 visit.
* Subjects who have a history of aspiration, or an underlying and/or a history of the symptoms that suggests high risks for aspiration by a investigator within 12 months before Day 1 (serious salivation requiring changing in a type of diet, chronic dysphagia that is difficult to swallow).
* Subjects who were treated with botulinum toxin for spasticity of upper limb less than 16 weeks before Day 1 visit.
* Subjects who underwent surgical interventions, phenol block, ethanol block or muscle afferent block (MAB) within 12 months before Day 1 visit, or these interventions are planned during the study period in any one of the finger (upper limb), wrist, elbow or shoulder muscles, which will be involved in the study.
* Subjects who placed a surgical cast or a dynamic splint within 3 months before Day 1 study visit, and/or these interventions are planned to be placed on the upper limb to be involved in the study.
* Subjects who were injected corticosteroid or an anesthetic agent into the finger (upper limb), wrist, or shoulder flexors, which will be involved in the study within 3 months before Day 1 visit, or these injections are planned during the study.
* Subjects who received constraint-induced movement therapy (CIMT) within 3 months before Day 1 visit or CIMT is planned during the blind phase.
* Subjects who underwent ultrasound therapy, transcutaneous electrical nerve stimulation (TENS) , electrical stimulation therapy, or acupuncture therapy in the upper arm, which will be involved in the study within 1 month before Day 1 visit, or these therapies are planned during the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- Japan (23):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokushima
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20343

REFERENCES:
- [Background] Abo M, Shigematsu T, Hara H, Matsuda Y, Nimura A, Yamashita Y, Takahashi K. Efficacy and Safety of OnabotulinumtoxinA 400 Units in Patients with Post-Stroke Upper Limb Spasticity: Final Report of a Randomized, Double-Blind, Placebo-Controlled Trial with an Open-Label Extension Phase. Toxins (Basel). 2020 Feb 18;12(2):127. doi: 10.3390/toxins12020127. PMID 32085529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 40 study centers in Japan, of which 38 centers enrolled participants.
Pre-assignment Details: A total of 131 participants were screened of which 7 participants were screen failures [reason being did not meet inclusion exclusion criteria (6) and withdrew consent (1)] and finally 124 participants were randomized (63 participants in the GSK1358820 240 units [U] group and 61 participants in the GSK1358820 400 U group).
Groups:
- GSK1358820 240 U: Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist (Flexor carpi radialis [B1], Flexor carpi ulnaris [B2]), finger (Flexor digitorum profundus [C1], Flexor digitorum superficialis [C2]), thumb (Flexor pollicis longus [D1], Adductor pollicis [D2]) and a single dose of matching placebo was injected into the muscles that acted on elbow flexors Biceps brachii [A1], Brachialis [A2], Brachioradialis [A3] during the double-blind phase. Participants who met the re-treatment criteria between Week 12 to 36 were treated with GSK1358820 400 U injections in the open-label phase (one injection each in Treatment cycles [cyc] 2, 3 and 4). Participants were re-treated up to 3 times with an interval of 12 weeks between treatments during the open-label phase.
- GSK1358820 400 U: Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist (Flexor carpi radialis [B1], Flexor carpi ulnaris [B2]), finger (Flexor digitorum profundus [C1], Flexor digitorum superficialis [C2]), thumb (Flexor pollicis longus [D1], Adductor pollicis [D2]) and a single dose of GSK1358820 160 U was injected into the muscles that acted on elbow flexors Biceps brachii [A1], Brachialis [A2], Brachioradialis [A3] during the double-blind phase. Participants who met the re-treatment criteria between Week 12 to 36 were treated with GSK1358820 400 U injections in the open-label phase (one injection each in Treatment cycles 2, 3 and 4). Participants were treated up to 3 times with an interval of 12 weeks between treatments during the open-label phase.
Period: Double Blind(Treatment cyc1,Upto Week48)
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Started | 63 | 61
Completed | 60 | 57
Not Completed | 3 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 3 | 1
Period: Open-label(Treatment cycle2,Upto Week48)
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Started (Participants who met retreatment criteria in Treatment cycle 1 and received second dose) | 60 | 57
Completed | 58 | 57
Not Completed | 2 | 0
Not completed — Protocol defined stopping criteria | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open-label(Treatment cycle3,Upto Week48)
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Started (Participants who met retreatment criteria in Treatment cycle 2 and received third dose) | 55 | 56
Completed | 54 | 55
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Open-label(Treatment cycle4,Upto Week48)
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Started (Participants who met retreatment criteria in Treatment cycle 3 and received fourth dose) | 43 | 40
Completed | 43 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1358820 240 U | GSK1358820 400 U | Total
Number analyzed (Participants) | 63 | 61 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (10.98) | 57.1 (9.90) | 57.2 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 53 | 46 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese/East Asian Heritage (AH)/South East AH | 63 | 60 | 123
  Asian & Native Hawaiian or other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Modified Ashworth Scale (MAS) Score Reduced at Least 1 From Baseline in the Elbow Flexors at Week 6
Description: MAS was used to measure the level of spasticity. The test was performed in a sitting position throughout the study. The affected parts were extended as fast as possible to grade the flexor muscle tones. It was scored on a scale of 0 to 4 as: 0=No increase in muscle tone, 1=Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension, 1+= Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half of ROM, 2 =More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved, 3= Considerable increase in muscle tone, passive movement difficult and 4= Affected part(s) rigid in flexion or extension. Higher scores= Worst outcome while lower scores= Better outcome.
Time Frame: Week 6
Population: Intent to treat 1 (ITT1) Population comprised of participants who were randomized in the study and who had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Percentage of participants | 50.8 | 68.9
Statistical Analysis 1: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Difference = 18.1, 95% CI 2-sided [1.1 to 35.0]

2. Secondary Outcome: Percentage of Participants Who Had MAS Score Reduction in Elbow, Wrist, Finger and Thumb Flexors up to Week 12
Description: MAS was used to measure the level of spasticity. The test was performed in a sitting position throughout the study. The affected parts were extended as fast as possible to grade the flexor muscle tones. It was scored on a scale of 0 to 4 as: 0=No increase in muscle tone, 1=Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension, 1+=Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM, 2=More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved, 3=Considerable increase in muscle tone, passive movement difficult and 4=Affected part(s) rigid in flexion or extension. Higher scores=worst outcome while lower scores=better outcome.
Time Frame: Week 2, Week 4, Week 6 and Week 12
Population: ITT1 Population. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles).
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Percentage of participants
  Elbow Flexion, Week 2, n=63,61 | 44.4 | 77.0
  Elbow Flexion, Week 4, n=63,61 | 52.4 | 73.8
  Elbow Flexion, Week 6, n=63,61 | 50.8 | 68.9
  Elbow Flexion, Week 12, n=63,61 | 33.3 | 45.9
  Wrist Flexion, Week 2, n=63,61 | 77.8 | 72.1
  Wrist Flexion, Week 4, n=63,61 | 82.5 | 73.8
  Wrist Flexion, Week 6, n=63,61 | 81.0 | 68.9
  Wrist flexion, Week 12, n=63,61 | 54.0 | 44.3
  Finger Flexion, Week 2, n=63,61 | 87.3 | 78.7
  Finger Flexion, Week 4, n=63,61 | 85.7 | 75.4
  Finger Flexion, Week 6, n=63,61 | 81.0 | 72.1
  Finger Flexion, Week 12, n =63,61 | 46.0 | 45.9
  Thumb Flexion, Week 2, n=60,54: number analyzed (Participants) | 60 | 54
  Thumb Flexion, Week 2, n=60,54 | 75.0 | 64.8
  Thumb Flexion, Week 4, n=60,54: number analyzed (Participants) | 60 | 54
  Thumb Flexion, Week 4, n=60,54 | 71.7 | 64.8
  Thumb Flexion, Week 6, n=60,54: number analyzed (Participants) | 60 | 54
  Thumb Flexion, Week 6, n=60,54 | 68.3 | 66.7
  Thumb flexion, Week 12,n=60,54: number analyzed (Participants) | 60 | 54
  Thumb flexion, Week 12,n=60,54 | 46.7 | 46.3
Statistical Analysis 1: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = 33.1, 95% CI 2-sided [17.0 to 49.2] — Week 2, Elbow flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 2: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = 21.7, 95% CI 2-sided [4.9 to 38.5] — Week 4, Elbow flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 3: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = 18.4, 95% CI 2-sided [1.3 to 35.5] — Week 6, Elbow flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 4: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = 12.9, 95% CI 2-sided [-4.2 to 30.1] — Week 12, Elbow flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 5: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -5.6, 95% CI 2-sided [-20.9 to 9.8] — Week 2, Wrist flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 6: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -8.6, 95% CI 2-sided [-23.0 to 5.9] — Week 4, Wrist flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 7: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -12.1, 95% CI 2-sided [-27.5 to 3.2] — Week 6, Wrist flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 8: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -9.6, 95% CI 2-sided [-27.2 to 7.9] — Week 12, Wrist flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 9: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -8.6, 95% CI 2-sided [-21.9 to 4.7] — Week 2, Finger flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 10: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -10.4, 95% CI 2-sided [-24.3 to 3.4] — Week 4, Finger flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 11: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -8.9, 95% CI 2-sided [-23.8 to 6.0] — Week 6, Finger flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 12: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -0.1, 95% CI 2-sided [-17.7 to 17.4] — Week 12, Finger flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 13: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -9.9, 95% CI 2-sided [-26.4 to 6.5] — Week 2, Thumb flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 14: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -6.7, 95% CI 2-sided [-23.6 to 10.3] — Week 4, Thumb flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 15: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -1.5, 95% CI 2-sided [-18.8 to 15.7] — Week 6, Thumb flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors
Statistical Analysis 16: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Adjusted rate difference = -0.5, 95% CI 2-sided [-18.8 to 17.9] — Week 12, Thumb flexion. Analysis was based on the Mantel-Haenszel method using Baseline MAS score of the elbow flexors

3. Secondary Outcome: Change From Baseline in MAS Scores in Elbow, Wrist, Finger and Thumb Flexors up to Week 12 (Mixed Model Repeated Measures [MMRM])
Description: The affected parts were extended as fast as possible to grade the flexor muscle tones. It was scored on a scale of 0 to 4 as: 0=No increase in muscle tone, 1=Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion/extension, 1+=Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM, 2=More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved, 3=Considerable increase in muscle tone, passive movement difficult and 4=Affected part(s) rigid in flexion/extension. Higher scores=worst outcome while lower scores=better outcome. Baseline was defined as the latest pre-first dose assessment with a non-missing value. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 2, Week 4, Week 6 and Week 12
Population: ITT1 Population. Only those participants with data available at the specified time points were analyzed (represented by n=x in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Scores on a scale
  Elbow Flexion, Week 2, n=63,60: number analyzed (Participants) | 63 | 60
  Elbow Flexion, Week 2, n=63,60 | -0.59 (0.089) | -1.07 (0.102)
  Elbow Flexion, Week 4, n=63,59: number analyzed (Participants) | 63 | 59
  Elbow Flexion, Week 4, n=63,59 | -0.7 (0.097) | -1.12 (0.110)
  Elbow Flexion, Week 6, n=63,59: number analyzed (Participants) | 63 | 59
  Elbow Flexion, Week 6, n=63,59 | -0.71 (0.107) | -1.09 (0.128)
  Elbow Flexion, Week 12, n=60,57: number analyzed (Participants) | 60 | 57
  Elbow Flexion, Week 12, n=60,57 | -0.35 (0.072) | -0.61 (0.101)
  Wrist Flexion, Week 2, n=63,60: number analyzed (Participants) | 63 | 60
  Wrist Flexion, Week 2, n=63,60 | -1.29 (0.120) | -1.21 (0.126)
  Wrist Flexion, Week 4, n=63,59: number analyzed (Participants) | 63 | 59
  Wrist Flexion, Week 4, n=63,59 | -1.45 (0.122) | -1.35 (0.132)
  Wrist Flexion, Week 6, n=63,59: number analyzed (Participants) | 63 | 59
  Wrist Flexion, Week 6, n=63,59 | -1.29 (0.115) | -1.31 (0.136)
  Wrist flexion, Week 12, n=60,57: number analyzed (Participants) | 60 | 57
  Wrist flexion, Week 12, n=60,57 | -0.69 (0.097) | -0.59 (0.107)
  Finger Flexion, Week 2, n=63,60: number analyzed (Participants) | 63 | 60
  Finger Flexion, Week 2, n=63,60 | -1.38 (0.113) | -1.28 (0.121)
  Finger Flexion, Week 4, n=63,59: number analyzed (Participants) | 63 | 59
  Finger Flexion, Week 4, n=63,59 | -1.49 (0.117) | -1.32 (0.130)
  Finger Flexion, Week 6, n=63,59: number analyzed (Participants) | 63 | 59
  Finger Flexion, Week 6, n=63,59 | -1.36 (0.118) | -1.22 (0.123)
  Finger Flexion, Week 12, n=60,57: number analyzed (Participants) | 60 | 57
  Finger Flexion, Week 12, n=60,57 | -0.63 (0.116) | -0.59 (0.097)
  Thumb Flexion, Week 2, n=60,53: number analyzed (Participants) | 60 | 53
  Thumb Flexion, Week 2, n=60,53 | -1.24 (0.123) | -0.96 (0.130)
  Thumb Flexion, Week 4, n=60,53: number analyzed (Participants) | 60 | 53
  Thumb Flexion, Week 4, n=60,53 | -1.29 (0.127) | -1.15 (0.138)
  Thumb Flexion, Week 6, n=60,53: number analyzed (Participants) | 60 | 53
  Thumb Flexion, Week 6, n=60,53 | -1.12 (0.119) | -1.10 (0.132)
  Thumb flexion, Week 12, n=57,51: number analyzed (Participants) | 57 | 51
  Thumb flexion, Week 12, n=57,51 | -0.69 (0.133) | -0.61 (0.144)
Statistical Analysis 1: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.75 to -0.22] — Week 2, Elbow flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 2: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.71 to -0.13] — Week 4, Elbow flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 3: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.71 to -0.04] — Week 6, Elbow flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 4: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.51 to -0.02] — Week 12, Elbow flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 5: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.27 to 0.42] — Week 2, Wrist flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 6: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.25 to 0.46] — Week 4, Wrist flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 7: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.37 to 0.33] — Week 6, Wrist flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 8: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.19 to 0.38] — Week 12, Wrist flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 9: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.23 to 0.43] — Week 2, Finger flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 10: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.17 to 0.52] — Week 4, Finger flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 11: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.20 to 0.48] — Week 6, Finger flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interaction, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 12: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.25 to 0.34] — Week 12, Finger flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interaction, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 13: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.28, 95% CI 2-sided [-0.08 to 0.63] — Week 2, Thumb flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 14: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.23 to 0.51] — Week 4, Thumb flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 15: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.33 to 0.38] — Week 6, Thumb flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 16: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.31 to 0.47] — Week 12, Thumb flexion. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects

4. Secondary Outcome: Change From Baseline in Principal Therapeutic Target of Disability Assessment Scale (DAS) - MMRM up to Week 12
Description: The investigator assessed 4 areas of disability namely hygiene, pain, dressing and limb posture and was graded using the 4-point DAS scale where (0=No functional disability, 1: Mild disability, 2: Moderate disability and 3=Severe disability). The investigator, in consultation with the participant, selected 1 functional disability item from the 4 areas of disability and assessed it as a principal therapeutic target. The maximum possible score was 3 where higher scores indicate severe disability and lowers scores indicate sound functional ability. Baseline value was defined as the latest pre-first dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 2, Week 4, Week 6 and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Scores on scale
  Week 2, n=63,60: number analyzed (Participants) | 63 | 60
  Week 2, n=63,60 | -0.34 (0.087) | -0.59 (0.085)
  Week 4, n=63,59: number analyzed (Participants) | 63 | 59
  Week 4, n=63,59 | -0.46 (0.096) | -0.62 (0.086)
  Week 6, n=63,59: number analyzed (Participants) | 63 | 59
  Week 6, n=63,59 | -0.52 (0.081) | -0.67 (0.078)
  Week 12, n=60,57: number analyzed (Participants) | 60 | 57
  Week 12, n=60,57 | -0.35 (0.082) | -0.63 (0.092)
Statistical Analysis 1: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.48 to 0.00] — Week 2. Analysis method was MMRM with Treatment, Visit, Treatment by visit interaction, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 2: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.42 to 0.09] — Week 4. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 3: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.37 to 0.08] — Week 6. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects
Statistical Analysis 4: Comparison: GSK1358820 240 U vs GSK1358820 400 U; Test type: Other; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.52 to -0.04] — Week 12. Analysis method was MMRM with Treatment, Visit, Treatment by visit interation, Baseline, and Baseline by visit interaction as fixed effects

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) After 84 Days of First Treatment
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment was categorized as SAE. Data for number of participants with any AE and any SAE is presented.
Time Frame: Up to 84 days post first treatment
Population: Safety1 Population. Safety1 Population comprised of all participants who were randomized in the study and who receive study treatment at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Participants
  Any AE | 29 | 31
  Any SAE | 4 | 5

6. Secondary Outcome: Number of Participants With AEs and SAEs-Overall Study Period
Description: as for outcome 5
Time Frame: Up to Week 48
Population: Safety1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Participants
  Any AE | 52 | 49
  Any SAE | 6 | 8

7. Secondary Outcome: Number of Participants With Abnormal Findings After Physical Examinations
Description: Physical examinations included assessment of lungs, cardiovascular system, and abdominal region (liver and spleen). This analysis was not planned and data was not collected and captured in the database.
Time Frame: Up to Week 48
Population: Safety1 Population. This analysis was not planned and data was not collected and captured in the database.
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Hematology parameters along with their normal ranges included: basophils (0 to 2 percent), eosinophils (0 to 8 percent), hemoglobin (135 to 175 grams/liter), hematocrit (0.397 to 0.524 proportion of red blood cells in blood), lymphocytes (18 to 49 percent), monocytes (2 to 10 percent), total neutrophils (40 to 75 percent), platelet count (140 to 340 giga cells/liter), red blood cell count (4.3 to 5.7 trillion cells/liter), white blood cell count (3.3 to 9 giga cells/liter), mean corpuscular volume (85 to 102 femtoliters), mean corpuscular hemoglobin (28 to 34 picograms) and reticulocyte count (0.004 to 0.019 percent/ratio). Shift in values relative to normal range as high and low have been presented for categories having non-zero values.
Time Frame: Up to Week 48
Population: Safety1 Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 62 | 59
Participants
  Eosinophils, To high | 7 | 3
  Hemoglobin, To low | 5 | 5
  Hemoglobin, To high | 1 | 5
  Hematocrit, To low | 5 | 5
  Hematocrit, To high | 4 | 6
  Lymphocytes, To low | 11 | 11
  Lymphocytes, To high | 0 | 1
  Mean corpuscle hemoglobin, To low | 2 | 1
  Mean corpuscle hemoglobin, To high | 1 | 3
  Mean corpuscle volume, To low | 3 | 0
  Mean corpuscle volume, To high | 1 | 2
  Monocytes, To high | 0 | 4
  Total neutrophils, To low | 0 | 1
  Total neutrophils, To high | 6 | 11
  Platelet count, To low | 2 | 1
  Platelet count, To high | 7 | 4
  Red blood cell count, To low | 2 | 2
  Red blood cell count, To high | 2 | 7
  Reticulocytes, To high | 4 | 5
  White blood cell count, To low | 0 | 1
  White blood cell count, To high | 3 | 3

9. Secondary Outcome: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Clinical chemistry parameters assessed were alkaline phosphatase (100 to 325 international units/liter), alanine amino transferase (5 to 45 international units/liter), aspartate amino transferase (10 to 40 international units/liter), direct bilirubin (0 to 3.42 micromoles/liter), total bilirubin (3.42 to 20.52 micromoles/liter), calcium (2.0958 - 2.5948 millimoles/liter), creatinine (53.924 - 91.936 micromoles/liter), potassium (3.5 - 5 millimoles/liter), sodium (137 - 147 millimoles/liter), total protein (67 - 83 grams/liter), urea/blood urea nitrogen (BUN) [2.856 - 7.14 millimoles/liter]. Shift in values relative to normal range as high and low have been presented for categories having non-zero values.
Time Frame: Up to Week 48
Population: Safety 1 Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 62 | 59
Participants
  Alkaline Phosphatase, High | 5 | 6
  Alanine amino transferase, High | 8 | 6
  Aspartate amino transferase, High | 3 | 2
  Direct bilirubin, High | 1 | 2
  Total bilirubin, High | 0 | 2
  Calcium, Low | 0 | 1
  Creatinine, Low | 5 | 1
  Creatinine, High | 3 | 2
  Potassium, Low | 1 | 1
  Potassium, High | 1 | 1
  Sodium, Low | 5 | 2
  Sodium, High | 1 | 0
  Total protein, Low | 11 | 14
  Total protein, High | 1 | 1
  Urea/BUN, Low | 2 | 3
  Urea/BUN, High | 7 | 5

10. Secondary Outcome: Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Analysis
Description: Urinalysis parameters assessed were urine occult blood, urine protein . In this dipstick test, occult blood and protein in urine samples were recorded as negative trace, 1+, 2+, and 3+ (the plus sign increases with occult blood or proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive etc). Number of participants with worst-case urinalysis results post-Baseline relative to Baseline by dipstick analysis have been presented.
Time Frame: Up to Week 48
Population: Safety 1 Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 61 | 59
Participants
  Occult blood, Any increase | 11 | 11
  Occult blood, Increase to trace | 4 | 2
  Occult blood, Increase to 1+ | 2 | 7
  Occult blood, Increase to 2+ | 1 | 2
  Occult blood, Increase to 3+ | 4 | 0
  Protein, Any increase | 9 | 14
  Protein, Increase to trace | 4 | 11
  Protein, Increase to 1+ | 4 | 2
  Protein, Increase to 2+ | 1 | 0
  Protein, Increase to 3+ | 0 | 1
  Protein, Increase to 4+ | 0 | 0

11. Secondary Outcome: Change From Baseline in Vital Sign Parameters Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 12 and Week 48
Description: Vital sign parameters SBP and DBP were measured in a semi-recumbent position after a 5-minute rest. If measurement in a semi-recumbent position was difficult, measurement in another position (e.g., sitting) was acceptable. The measurement was performed always in the same position during the study period. SBP and DBP were measured using an automated device. Baseline value was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 12 and Week 48
Population: Safety1 Population. Only those participants with data available at the indicated time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Millimeters of mercury
  SBP, Week 12; n=60, 57: number analyzed (Participants) | 60 | 57
  SBP, Week 12; n=60, 57 | 0.8 (11.29) | 1.3 (11.19)
  DBP, Week 12; n=60, 57: number analyzed (Participants) | 60 | 57
  DBP, Week 12; n=60, 57 | 0.5 (8.01) | 0.1 (10.39)
  SBP, Week 48; n=57, 56: number analyzed (Participants) | 57 | 56
  SBP, Week 48; n=57, 56 | -1.6 (13.85) | -1.7 (14.60)
  DBP, Week 48; n=57, 56: number analyzed (Participants) | 57 | 56
  DBP, Week 48; n=57, 56 | -1.8 (10.01) | -1.2 (11.42)

12. Secondary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate at Week 12 and Week 48
Description: Vital sign parameter heart rate was measured in a semi-recumbent position after a 5-minute rest. If measurement in a semi-recumbent position was difficult, measurement in another position (e.g., sitting) was acceptable. The measurement was performed always in the same position during the study period. Heart rate was measured using an automated device. Baseline value was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 12 and Week 48
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Beats per minute
  Week 12; n=60, 57: number analyzed (Participants) | 60 | 57
  Week 12; n=60, 57 | 0.2 (9.95) | 2.6 (8.20)
  Week 48; n=57, 56: number analyzed (Participants) | 57 | 56
  Week 48; n=57, 56 | 0.5 (10.05) | -0.1 (9.01)

13. Secondary Outcome: Change From Baseline in Vital Sign Parameter Temperature at Week 12 and Week 48
Description: Vital sign parameter temperature was measured orally, intra-aurally, or axillary fossa, the participant was instructed to refrain from eating food or drinking beverage within 5 minutes before the measurement. The method for the measurement of body temperature was same throughout the study. Baseline value was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 12 and Week 48
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | GSK1358820 240 U | GSK1358820 400 U
Number analyzed (Participants) | 63 | 61
Degree Celsius
  Week 12; n=59, 56: number analyzed (Participants) | 59 | 56
  Week 12; n=59, 56 | -0.03 (0.428) | -0.08 (0.466)
  Week 48; n=57, 56: number analyzed (Participants) | 57 | 56
  Week 48; n=57, 56 | 0.00 (0.505) | -0.06 (0.461)

ADVERSE EVENTS:
Time Frame: Non-serious AE and SAE were collected from start of the study drug until Week 48 in double blind-phase (Treatment cycle1) and from day of injection in Treatment cycles 2, 3 and 4 until Week 48 (48 weeks after first treatment) for participants in the respective treatment cycles in Open-label phase.
Description: Safety1 Population was used for assessment of nSAE and SAE during double-blind (Treatment Cycle 1). Safety2, Safety3 and Safety4 Population were used for assessment of nSAEs and SAEs during Treatment Cycles 2, 3 and 4, respectively. All participants received GSK1358820 400 U in open-label phase (Treatment Cycles 2, 3 and 4).
Groups:
- GSK1358820 240 U (Double Blind-Treatment Cycle 1): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and matching placebo was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase.
- GSK1358820 400 U (Double Blind-Treatment Cycle 1): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and GSK1358820 160 U was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase.
- GSK1358820 240 U (Open Label-Treatment Cycle 2): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and matching placebo was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase. Participants who met the eligibility criteria for re-treatment between Week 12 to Week 36 were treated with GSK1358820 400 U injection in the open-label phase (Treatment cycle 2).
- GSK1358820 400 U (Open labelTreatment Cycle 2): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and GSK1358820 160 U was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase. Participants who met the eligibility criteria for re-treatment between Week 12 to Week 36 were treated with GSK1358820 400 U injection in the open-label phase (Treatment cycle 2).
- GSK1358820 240 U (Open Label-Treatment Cycle 3): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and matching placebo was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase. Participants who met the eligibility criteria for re-treatment between Week 12 to Week 36 were treated with GSK1358820 400 U injections in Treatment cycle 2 and 3 of open-label phase with an interval of 12 weeks between treatments.
- GSK1358820 400 U (Open Label-Treatment Cycle 3): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and GSK1358820 160 U was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase. Participants who met the eligibility criteria for re-treatment between Week 12 to Week 36 were treated with GSK1358820 400 U injections in Treatment cycles 2 and 3 of open-label phase with an interval of 12 weeks between treatments.
- GSK1358820 240 U (Open Label-Treatment Cycle 4): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and matching placebo was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase. Participants who met the eligibility criteria for re-treatment between Week 12 to Week 36 were treated with GSK1358820 400 U injections in Treatment cycle 2, 3 and 4 of open-label phase with an interval of 12 weeks between treatments.
- GSK1358820 400 U (Open Label-Treatment Cycle 4): Participants were injected with a single dose of GSK1358820 240 U into the muscles that act on the wrist and GSK1358820 160 U was injected into the muscles that acted on elbow flexors on Day 1 during the double-blind phase. Participants who met the eligibility criteria for re-treatment between Week 12 to Week 36 were treated with GSK1358820 400 U injections in Treatment cycles 2, 3 and 4 of open-label phase with an interval of 12 weeks between treatments.
Arm/Group | GSK1358820 240 U (Double Blind-Treatment Cycle 1) | GSK1358820 400 U (Double Blind-Treatment Cycle 1) | GSK1358820 240 U (Open Label-Treatment Cycle 2) | GSK1358820 400 U (Open labelTreatment Cycle 2) | GSK1358820 240 U (Open Label-Treatment Cycle 3) | GSK1358820 400 U (Open Label-Treatment Cycle 3) | GSK1358820 240 U (Open Label-Treatment Cycle 4) | GSK1358820 400 U (Open Label-Treatment Cycle 4)
All-Cause Mortality (participants affected / at risk) | 0/63 | 1/61 | 0/60 | 0/57 | 0/55 | 0/56 | 0/43 | 0/40
Serious Adverse Events (participants affected / at risk) | 4/63 | 5/61 | 1/60 | 2/57 | 2/55 | 1/56 | 0/43 | 2/40
Other Adverse Events (participants affected / at risk) | 19/63 | 24/61 | 7/60 | 11/57 | 12/55 | 6/56 | 7/43 | 13/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1358820 240 U (Double Blind-Treatment Cycle 1) (N=63) | GSK1358820 400 U (Double Blind-Treatment Cycle 1) (N=61) | GSK1358820 240 U (Open Label-Treatment Cycle 2) (N=60) | GSK1358820 400 U (Open labelTreatment Cycle 2) (N=57) | GSK1358820 240 U (Open Label-Treatment Cycle 3) (N=55) | GSK1358820 400 U (Open Label-Treatment Cycle 3) (N=56) | GSK1358820 240 U (Open Label-Treatment Cycle 4) (N=43) | GSK1358820 400 U (Open Label-Treatment Cycle 4) (N=40)
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Decreased activity (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1358820 240 U (Double Blind-Treatment Cycle 1) (N=63) | GSK1358820 400 U (Double Blind-Treatment Cycle 1) (N=61) | GSK1358820 240 U (Open Label-Treatment Cycle 2) (N=60) | GSK1358820 400 U (Open labelTreatment Cycle 2) (N=57) | GSK1358820 240 U (Open Label-Treatment Cycle 3) (N=55) | GSK1358820 400 U (Open Label-Treatment Cycle 3) (N=56) | GSK1358820 240 U (Open Label-Treatment Cycle 4) (N=43) | GSK1358820 400 U (Open Label-Treatment Cycle 4) (N=40)
Nasopharyngitis (Infections and infestations) | 11 | 7 | 2 | 1 | 4 | 0 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 7 | 4 | 5 | 3 | 3 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 4 | 3 | 3 | 1 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 2 | 3 | 0 | 0 | 2 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT03261167/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT03261167/SAP_001.pdf